CLINICAL TRIAL: NCT00753779
Title: Efficacy of WelChol® as an Add-on to Simvastatin Therapy
Brief Title: A Study to Determine the Effect of WelChol Tablets on Cholesterol in Patients Who Have Been Taking Simvastatin for at Least 4 Weeks.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Senior Director Metobolic Research, Daiichi Sankyo, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WEL-405
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): colesevelam HCl Tablets and simvastatin tablets
  Interventions: Drug: colesevelam HCl tablets, and simvastatin tablets
- 2 (Placebo Comparator): simvastatin and Welchol placebo
  Interventions: Drug: simvastatin tablets and colesevelam HCl placebo

INTERVENTIONS:
Drug: colesevelam HCl tablets, and simvastatin tablets — colesevelam HCl tablets, 6/day simvastatin tablet, 1/day
  Arms: 1
Drug: simvastatin tablets and colesevelam HCl placebo — simvastatin tablet, 1/day; Welchol placebo tablets, 6/day
  Arms: 2

SUMMARY:
The primary objective is to determine the effect of WelChol tablets on serum lipids, lipoproteins, apolipoproteins, and lipoprotein particle size in patients who were stabilized on simvastatin therapy for at least 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* > or = to 18 years of age
* On a stable dose of simvastatin for 4 or more weeks
* LDL-C > or = to 115 mg/dL and < or = to 250 mg/dL
* TG < 300 mg/dL
* Women are not pregnant or breast-feeding or planning to become pregnant
* Women had a hysterectomy or tubal ligation or are post menopausal or are practicing an acceptable method of contraception

Exclusion Criteria:

* BMI > 40
* Allergic to colesevelam HCl
* History of swallowing disorder
* History of gastrointestinal motility disorder
* Any disorder that might interfere with the study
* History of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2002-11; Primary Completion 2003-06 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
The percent change in LDL-C from baseline to endpoint | 6 weeks

SECONDARY OUTCOMES:
The absolute change in LDL-C from baseline to endpoint | 6 weeks
The absolute and % change of total cholesterol | 6 Weeks
The absolute and % change in triglycerides | 6 Weeks
The absolute and % change in HDL-C | 6 Weeks

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Los Angeles, California
  - Castle Rock, Colorado
  - Jacksonville, Florida
  - Pembroke Pines, Florida
  - St. Petersburg, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Rochester, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Bartlett, Tennessee
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington